CLINICAL TRIAL: NCT04043273
Title: Treatment-related Benefit and Satisfaction in Fabry Patients. Insight in Patients Expectations and Preferences (SATIS-Fab)
Brief Title: Treatment-related Benefit and Satisfaction in Fabry Patients. Insight in Patients Expectations and Preferences
Status: Completed | Type: Observational
Sponsor: Amicus Therapeutics France SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: SATIS-Fab
Record Dates: First submitted 2019-06-28; First posted 2019-08-02 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Fabry Disease; Anderson Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Whole cohort: The whole cohort will be divided into clusters according to patients expectations and preferences regarding their treatment
  Interventions: Behavioral: Noninterventional characterization of patients expectations and preferences regarding their treatment

INTERVENTIONS:
Behavioral: Noninterventional characterization of patients expectations and preferences regarding their treatment — Patients will be clustered before and after a principal components analysis (PCA) on Patients Needs Questionnaire (PNQ). Observations will be clustered by the Ward method. The number of clusters will be chosen using the Kolinski criteria. Characteristics of patients will be described by cluster.

SUMMARY:
In the shared decision-making process, patients should express their expectations and preferences regarding treatment to the physician. A specific questionnaire addressing needs and expectations of Fabry patients has been built at the initiative of Amicus. In addition, this questionnaire also evaluates the benefit of treatment from the patient's perspective. Nothing is known until now on patient's expectations, potential clustering of patients regarding their expectations and evaluation of treatment benefit from the patients perspective.

Study objectives are differentiated according to the study phase (inclusion and follow-up). At inclusion, the primary objective is to cluster patients according to their needs and expectations regarding treatment. During follow-up, the primary objective is to evaluate treatment benefit in relation with patients needs and expectations.

DETAILED DESCRIPTION:
Prospective, longitudinal, non-comparative, open-label, multicentre, non interventional cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 16 years old
* Diagnosed with Fabry disease
* With amenable mutation
* Decision by clinician to start or pursue ongoing ERT or migalastat
* Non-opposition form to participate in the study signed

Exclusion Criteria:

- Concomitant patient participation in an interventional clinical study (Category 1 interventional research or category 2 interventional research according to the Jardé law classification in France)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Fabry disease with the potential to be treated either by ERT or migalastat in real-life conditions and according to the SmPC
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Homogeneous clusters of patients according to their needs and expectations towards the treatment received. | Baseline
  Number of clusters will be defined using a non-supervised classification method.
Treatment benefit, derived from Patients Benefit Index (PBI), in relation to patients needs and expectations towards their specific treatment. | 12 month
  Patients Benefit Index (PBI): descriptive statistics. The PBI will be calculated by reference to the PNQ measured at the preceding visit
  The proportion of patients with PBI ≥ 1 will be described with a two-sided 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lidove, MD, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (15):
- France (15):
  - CHU d'Angers, Angers
  - CHU Pellegrin, Bordeaux
  - Hôpital Côte de Nacre, Caen
  - CHU de Dijon, Dijon
  - CHRU de Lille, Lille
  - Hôpital Femme Mère Enfant, Lyon
  - Hôpital de la Conception, Marseille
  - CHU de Nantes, Nantes
  - Hopital Tenon, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No